CLINICAL TRIAL: NCT06200441
Title: Correlation of Serum Gasdermin-D and NLRP-3 Inflammasome Levels With GVHD Biomarkers and Endothelial Damage Markers in Graft-Versus-Host Disease in AML Patients Undergoing Allogeneic Bone Marrow Transplantation
Brief Title: Correlation of Serum Gasdermin-D and NLRP-3 Inflammasome Levels With GVHD Biomarkers and Endothelial Damage Markers in Graft-Versus-Host Disease
Status: Withdrawn | Type: Observational
Why Stopped: Kits were not available due to lack of sponsorship
Sponsor: Ugur Arzu Kulu (Other)
Responsible Party: Sponsor-Investigator, Ugur Arzu Kulu, Research Assistant, Ankara University
Organization: Ankara University (Other)
Other Study IDs: AnkaraUniversityMedicine
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia, Adult; Graft Versus Host Disease; Endothelial Dysfunction
Keywords: Acute Myeloid Leukemia, Adult; Graft Versus Host Disease; Pyroptotic Cell Death; Gasdermin-D; NLR Family, Pyrin Domain-Containing 3 Protein; Endothelial Dysfunction
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Developing GVHD: Group of patients who developed GVHD during follow-up in patients who underwent allogeneic hematopoteic stem cell transplantation for AML
- non-GVHD: Group of patients who did not develop GVHD during follow-up in patients who received allogeneic hematopoteic stem cell transplantation for AML

SUMMARY:
The investigators aimed to reveal the relationship between serum markers of pyroptosis, GVHD biomarkers and endothelial damage markers in patients who were planned for allogeneic stem cell transplantation for AML and developed GVHD during follow-up. Secondary outcomes of the study were to demonstrate the role of pyroptosis in the pathophysiology of GVHD and transplantation-associated endothelial injury using serum plasma samples; the efficacy of GVHD biomarkers used to demonstrate organ-specific involvement; and the efficacy of GVHD biomarkers and endothelial injury markers in predicting the development of GVHD, transplantation-associated endothelial injury and non-relapse mortality.

DETAILED DESCRIPTION:
In the study, in patients who were planned to receive allogeneic stem cell transplantation for AML, pre-transplant period (before and after central catheter insertion) and post-transplant period (+1, +7, +14, +28, +60 and +100 days in the post-transplant period) serum pyroptosis markers (Serum Gasdermin-D and NLRP-3 Inflammasome levels), GVHD biomarkers (REG-3 alpha, ST2, ELAFIN, HGF, ILR2-alpha, CXCL 9, CXCL 10, CXCL11, BAFF, TNF-alpha, I IL8, IL6 , IL18 , I IL1-beta , IL12 , IFN-gamma) and endothelial damage markers (serums-ICAM , sE-selectin , sVCAM , ANG2 , CRP , vWF , Factor 8 , LDH , d-dimer , transaminase enzyme levels and before transplantation, The aim of this study was to determine the relationship between basic biomarkers in pyroptosis and biomarkers with high predictive value in GVHD and markers of endothelial damage in patients who develop GVHD during follow-up using nail bed capillaroscopic examination and fibroelastographic evaluation to be performed on the twenty-first and hundredth days after transplantation.The serum samples obtained will be compared with the groups of patients with and without GVHD at the planned 1-year follow-up.

Patients diagnosed with AML between 15.11.2023 and 15.11.2024 will be included in the study and a total of 2 years of clinical follow-up is planned.

In case of loss of participants during follow-up, the study planned to recruit new patients with AML who were scheduled for transplantation between November 15, 2023 and November 15, 2024.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with acute myeloid leukemia undergoing allogeneic bone marrow transplantation
* Patients followed up by the Department of Hematology, Ankara University Faculty of Medicine Hospitals

Exclusion Criteria:

* Patients under 18 years of age
* Patients with non-AML transplant indication
* Patients not followed up by the Department of Hematology, Ankara University Faculty of Medicine Hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who underwent allogeneic hematopoteic stem cell transplantation for AML and were followed up by Ankara University Hematology Department
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
The relationship between pyroptosis, GVHD and endothelial damage in allogeneic bone marrow transplant patients | The pre- and post-transplant serum samples,capillaroscopic and fibroelastographic examinations will be performed for each participant at the specified time interval until post-transplant 100th day
  To reveal the relationship between basic biomarkers in pyroptosis and biomarkers with high predictive value in GVHD and endothelial damage markers in AML (acute myeloid leukemia) patients with allogeneic bone marrow transplantation

SECONDARY OUTCOMES:
Efficacy of used GVHD biomarkers in indicating organ-specific involvement | The pre- and post-transplant serum samples,capillaroscopic and fibroelastographic examinations will be performed for each participant at the specified time interval until post-transplant 100th day
  Effect of REG-3 alpha, ELAFIN and HGFs in demonstrating organ specificity in GVHD development
The effectiveness of biomarkers in predicting the development of GVHD, transplant-related endothelial injury, and non-relapse mortality | The pre- and post-transplant serum samples,capillaroscopic and fibroelastographic examinations will be performed for each participant at the specified time interval until post-transplant 100th day
  The effectiveness of the biomarkers in predicting the development of GVHD, transplantation-related endothelial damage, and non-relapse mortality in the planned one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Kurt Yüksel, Study Director — Ankara University, Department of Hematology
Locations (1):
- Ankara University, Department of Hematology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No